CLINICAL TRIAL: NCT01666600
Title: A Phase I/II, Randomized, Open-label, Multi-centre Study of BIBF1120 + Reirradiation (R-RT) Versus Reirradiation in the Treatment of Patients With First or Second Progression of Glioblastoma
Brief Title: NOA-12: BIBF1120 and R-RT in Glioblastoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Interim Analysis for Feasibility
Sponsor: Prof. Dr. Wolfgang Wick (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Wolfgang Wick, Professor Dr. med., University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NONK-3/NOA-12
Record Dates: First submitted 2012-07-12; First posted 2012-08-16 (Estimated); Last update posted 2017-11-01 (Actual); Status verified 2017-10

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma | interventions — nintedanib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIBF 1120 + reirradiation (Experimental): 2 x minimal tolerated dose BIBF 1120 per day in combination with radiotherapy (2 Gy / fraction; 36 Gy in total)
  Interventions: Drug: BIBF 1120
- reirradiation alone (Active Comparator): radiotherapy (2 Gy / fraction; 36 Gy in total)
  Interventions: Radiation: radiotherapy

INTERVENTIONS:
Drug: BIBF 1120 — BIBF 1120 is given as 2 x minimal tolerated dose per day as long as as a clinical benefit is considered by the treating physician.
  Arms: BIBF 1120 + reirradiation
Radiation: radiotherapy — 36 Gy, 2 Gy / fraction, 18 fractions
  Arms: reirradiation alone

SUMMARY:
Patients with glioblastoma at first or second progression who have failed standard treatment that must have included radiochemotherapy with temozolomide and who are a candidate for a reirradiation can be included into the trial. In the phase I part the minimal tolerated dose (MTD)of BIBF 1120 in combination with radiotherapy will be investigated. Subjects in phase II will be randomised to receive reirradiation alone or reirradiation + 2 x MTD BIBF1120.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients with a recurrence / progression of glioblastoma either not being eligible for tumour resection or having macroscopic residual tumour after resection of the recurrence
* Diagnosis of glioblastoma must be proven histologically and progress must be documented by MRI. MRI images must not be older than 2 weeks before first dosing/start of RT
* Not more than two prior therapy regimens including one or two resections, one or two chemotherapies (one temozolomide containing concomitant to radiotherapy) and one radiotherapy (RT) for the brain tumour
* Previous irradiation therapy of the primary tumour with a maximal dose of 60 Gy; at least 8 months since the end of preirradiation
* Candidate for reirradiation with recurrent tumour visible on MRIT1 (Gd) and with the largest diameter measuring 1 cm to 5 cm
* Informed consent
* Age ≥ 18 years, smoking or non-smoking, of any ethnic origin
* Karnofsky performance index (KPI) ≥ 60%
* Neutrophile counts > 1500/μl / Platelet counts > 80.000/μl /Haemoglobin > 10 g/dl / Serum creatinine < 1.5-fold upper normal range / Bilirubin, AST or ALT < 2,5-fold upper normal range unless attributed to anticonvulsants / Alkaline phosphatase < 2,5-fold upper normal range
* Adequate contraception
* If on steroids, stable or decreasing treatment with steroids within 5 days before treatment start

Exclusion Criteria:

* More than one RT of brain, prior first radiotherapy with more than 60 Gy
* Cumulative total dose on the optical chiasm >54 Gy for 2 Gy/fraction, α/β=2
* Prior treatment with bevacizumab, iodine seeds and/or brachytherapy
* Unable to undergo MRI
* Past medical history of diseases with poor prognosis according to the judgement of the Investigator, e.g. severe coronary heart disease, severe diabetes, immune deficiency, residual deficits after stroke, severe mental retardation
* HIV or hepatitis infection
* Pregnancy or breast feeding
* Treatment within any other clinical trial parallel to the treatment phase of the current study or within 30 days before inclusion
* Known coronary artery disease, significant cardiac arrhythmias or severe congestive heart failure (NYHA class III - IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2012-08; Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Maximal tolerated dose of BIBF 1120 in combination with reirradiation (Phase I) | day 0, 8, 15 and 17 post-dose during phase I

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability of BIBF1120 | Up to 90 days follow-up
Progression-free survival | Time from randomization until death or disease progression
Objective response rates (OR) | Time from randomization until response
Overall survival | Time from randomization until death
Quality of life as determined by EORTC QLQ-C15 PAL and the EORTC brain module QLQ-BN 20 | Screening and 6-weekly after radiotherapy
Cognitive function determined by MMSE | Screening and 6-weekly after end of radiotherapy

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Heidelberg, Department of Neurooncology, Heidelberg, Baden-Wurttemberg
  - University Hospital Heidelberg, Department of Pharmacology, Heidelberg, Baden-Wurttemberg